CLINICAL TRIAL: NCT01199393
Title: Genetic Polymorphisms Predict Chemotherapeutic Outcomes in Patients With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director, Peking University Cancer Hospital & Institute
Other Study IDs: snp
Record Dates: First submitted 2010-08-31; First posted 2010-09-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasm; Drug Therapy; Polymorphism,Single Nucleotide
Keywords: breast neoplasm; drug therapy; polymorphism; gene
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — about 4ml peripheral vein blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators want to research whether genetic polymorphisms of drug-metabolizing enzymes can be used to predict chemotherapeutic outcomes in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
1. Patients evaluation On all patients a complete clinical history and physical examination is performed, including routine hematology and biochemistry analyses. Hematology and biochemistry analyses are repeated at the end of each cycle. Toxicity is classified according to WHO criteria at each cycle for each patient. Response is assessed after two cycles of chemotherapy and every two cycles thereafter, using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines.
2. Sample collection and SNP genotyping Venous blood (4 ml) is collected from each subject and placed into tubes containing EDTA. Genomic DNA is isolated with a DNA Blood isolation kit.Genotypes are performed by PCR-RFLP, PCR-DHPLC and PCR-direct sequencing, etc.
3. Statistical Analysis x2 test is used to summarize the association of response and adverse events to chemotherapy with genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer
* Female
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* At least one measurable lesion
* Normal cardiac, hepatic, renal and bone marrow functions
* Life expectancy ≥3 months
* Discontinuity of previous chemotherapy for a minimum of 4 weeks

Exclusion Criteria:

* Central nervous system metastases
* Serious or uncontrolled concurrent medical illness
* History of other malignancies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Response to chemotherapy | 6 months
  Response to chemotherapy is evaluated by Response Evaluation Criteria in Solid Tumors(RESIST).

SECONDARY OUTCOMES:
Time to disease progression | 1 year
  Time to disease progression is measured from the date therapy is initiated to the date of documented disease progression.
Overall survival | 5 years
  Overall survival is measured from the date therapy is initiated to the date of death or final follow-up.
Toxicity | 6 months
  Toxicity, as a measure of safety and tolerability, is assessed by the percent of participants with adverse events according to National Cancer Institute Common Toxicity Criteria (NCI-CTC). Possible toxicities include neutropenia, anemia, thrombocytopenia, nausea and vomitting, allergy, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Ningning Dong, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Jun Jia, MD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China